CLINICAL TRIAL: NCT00707993
Title: A Multicenter, Randomized, Double-Blind Study to Evaluate the Efficacy and Safety of Alogliptin Compared to Glipizide in Elderly Subjects With Type 2 Diabetes
Brief Title: Efficacy and Safety of Alogliptin Compared to Glipizide in Elderly Diabetics
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYR-322_303; 2008-000959-10 (Registry Identifier: EudraCT); U1111-1112-7905 (Registry Identifier: WHO)
Record Dates: First submitted 2008-06-27; First posted 2008-07-02 (Estimated); Results first posted 2013-05-24 (Estimated); Last update posted 2013-05-24 (Estimated); Status verified 2013-05

CONDITIONS: Diabetes Mellitus
Keywords: Glucose Metabolism Disorder; Dysmetabolic Syndrome; Type II Diabetes; Diabetes Mellitus; Lipoatrophic; Dyslipidemia; Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus; Glucose Metabolism Disorders; Diabetes Mellitus, Type 2; Dyslipidemias | interventions — alogliptin; Glipizide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alogliptin 25 mg QD (Experimental)
  Interventions: Drug: Alogliptin
- Glipizide 5 mg QD (Active Comparator)
  Interventions: Drug: Glipizide

INTERVENTIONS:
Drug: Alogliptin — Alogliptin 25 mg, tablets, orally, once daily and glipizide placebo matching tablets, orally, once daily for up to 52 weeks.
  Other Names: SYR110322; SYR-322
  Arms: Alogliptin 25 mg QD
Drug: Glipizide — Alogliptin placebo-matching tablets, orally, once daily and glipizide 5 mg to 10 mg, tablets, orally, once daily up to 52 weeks.
  Other Names: Glucotrol
  Arms: Glipizide 5 mg QD

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of alogliptin, once daily (QD), compared to glipizide in elderly diabetic patients who have not received treatment or are on a single oral medication.

DETAILED DESCRIPTION:
Type 2 diabetes is among the most common chronic condition in adults 65 years of age or older. A recent National Health and Nutrition Examination Survey reported that more than 20% of adults aged 65 years or older have diabetes. These individuals are often under-treated with respect to glucose-lowering medications, and their care is complicated by the extent of their clinical and functional status. Age-related changes in physiology, diabetes-associated illnesses and other illnesses (such as renal, cardiac, and hepatic insufficiency), as well as use of multiple medications make standard oral anti-hyperglycemic therapy and insulin use problematic. In addition, hypoglycemia is more common and severe in older rather than younger patients taking oral antidiabetic drugs which can precipitate serious events such as falls and hip fractures. While avoidance of hypoglycemia is paramount in elderly diabetic patients, many commonly used medications are associated with a substantial risk for hypoglycemia. New classes of drug which avoid such complications in the elderly population are of increasing interest as this population continues to expand.

Takeda is developing SYR-322 (alogliptin) for the improvement of glycemic control in patients with type 2 diabetes mellitus. Alogliptin is an inhibitor of the dipeptidyl peptidase IV enzyme. Dipeptidyl peptidase IV is thought to be primarily responsible for the degradation of 2 peptide hormones released in response to nutrient ingestion. It is expected that inhibition of dipeptidyl peptidase IV will improve glycemic (glucose) control in patients with type 2 diabetes.

This study will compare the effectiveness and safety of alogliptin with that of glipizide (a commonly used diabetes medication) in adults who are 65 to 90 years of age with Type 2 diabetes. Individuals who participate in this study will either have failed diet and exercise therapy alone during the 2 months before Screening, or will have been receiving a single oral antidiabetic medication without obtaining good blood glucose (sugar) control.

Each participant will be required to commit to screening visits. Study participation is anticipated to be up to 59 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of type 2 diabetes mellitus with either:

  * Failed diet and exercise therapy alone as demonstrated by inadequate glycemic control while receiving no antidiabetic treatment within the two months prior to Screening, or
  * Failed treatment with oral monotherapy alone (may include treatment with two or more antidiabetic agents if for less than 7 days) as demonstrated by inadequate glycemic control within the two months prior to Screening.
* Body mass index greater than or equal to 23 kg/m2 and less than or equal to 45 kg/m2.
* If regularly using other, non-excluded medications, must be on a stable dose for at least the 4 weeks prior to Screening.
* Females of childbearing potential who are sexually active must agree to use a medically accepted means of contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.
* Able and willing to monitor their own blood glucose concentrations with a home glucose monitor.
* No major illness or debility that in the investigator's opinion prohibits the participant from completing the study.

Exclusion Criteria:

* Systolic blood pressure greater than or equal to 160 mm Hg and/or diastolic pressure greater than or equal to 100 mm Hg.
* Hemoglobin less than or equal to 12 g/dL for males or less than or equal to 10 g/dL for females.
* Alanine aminotransferase greater than or equal to 3 times the upper limit of normal.
* Calculated creatinine clearance less than or equal to 50 mL/min.
* Thyroid-stimulating hormone level outside of the normal range.
* History of cancer, other than squamous cell or basal cell carcinoma of the skin, that has not been in full remission for at least 5 years prior to Screening.
* History of laser treatment for proliferative diabetic retinopathy within the 6 months prior to Screening.
* History of treated diabetic gastroparesis, gastric banding, or gastric bypass surgery.
* New York Heart Association Class III or IV heart failure regardless of therapy.
* History of coronary angioplasty, coronary stent placement, coronary bypass surgery, or myocardial infarction within the 6 months prior to Screening.
* History of any hemoglobinopathy that may affect determination of glycosylated hemoglobin.
* History of infection with Human Immunodeficiency Virus.
* History of a psychiatric disorder that will affect the participant's ability to participate in the study.
* History of angioedema in association with use of angiotensin-converting enzyme inhibitors or angiotensin-II receptor inhibitors.
* History of alcohol or substance abuse within the 2 years prior to Screening.
* History of treatment with any weight-loss drugs or oral or systemically injected glucocorticoids within the 3 months prior to Screening.
* Receipt of any investigational drug within the 30 days prior to Screening.
* Prior treatment in an investigational study of alogliptin.
* Clinically significant medical abnormality or disease or clinically significant abnormal findings at Screening (other than type 2 diabetes) that, in the opinion of the investigator, should exclude the participant from the study.
* Has donated more than 400 mL of blood within the 90 days preceding their participation in the study.
* Has hypersensitivity or has had an anaphylactic reaction(s) to any DPP-4 inhibitor drug.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 441 (Actual)
Dates: Start 2008-06; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: VP Biological Sciences, Study Director — Takeda
Locations (80):
- United States (36):
  - Alexander City, Alabama
  - Foothill Ranch, California
  - Huntington Park, California
  - Long Beach, California
  - Los Angeles, California
  - Redlands, California
  - Prospect, Connecticut
  - Bradenton, Florida
  - Fort Myers, Florida
  - Miami, Florida
  - Ormond Beach, Florida
  - Winter Park, Florida
  - Roswell, Georgia
  - Aurora, Illinois
  - La Porte, Indiana
  - South Bend, Indiana
  - Salisbury, Maryland
  - Clarkston, Michigan
  - Omaha, Nebraska
  - Hamilton, New Jersey
  - Albuquerque, New Mexico
  - Beachwood, Ohio
  - Westlake, Ohio
  - Zanesville, Ohio
  - Bensalem, Pennsylvania
  - Aiken, South Carolina
  - Greenville, South Carolina
  - Greer, South Carolina
  - Taylors, South Carolina
  - Corpus Christi, Texas
  - Dallas, Texas
  - Pasadena, Texas
  - San Antonio, Texas
  - Tomball, Texas
  - Ogden, Utah
  - Salt Lake City, Utah
- Hungary (3):
  - Budapest
  - Miskoic
  - Nyíregyháza
- India (4):
  - Karnāl, Haryana
  - Bangalore, Karnataka
  - Belagavi, Karnataka
  - Mumbai, Maharashrta
- Israel (6):
  - Ashkelon
  - Haifa
  - Holon
  - Nahariya
  - Rishon LeZiyyon
  - Safed
- Mexico (9):
  - Aguascalientes, Aguascalientes
  - Saltillo, Coahuila
  - Durango, Durango
  - Pachuca, Hidalgo
  - Morelia, Michoacán
  - Monterrey, Nuevo León
  - Guadalajara
  - Mexico City
  - Nezahualcóyotl
- Peru (3):
  - Arequipa
  - Lima
  - Piura
- Poland (3):
  - Gdansk
  - Krakow
  - Warsaw
- Romania (5):
  - Baia Mare
  - Brasov
  - Bucharest
  - Galati
  - Satu Mare
- Russia (3):
  - Arkhangelsk
  - Irkutsk
  - Smolensk
- South Africa (6):
  - Cape Town
  - Centurion
  - Durban
  - Johannesburg
  - Port Elizabeth
  - Pretoria
- Ukraine (2):
  - Donetsk
  - Kharkiv

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled at 110 investigative sites in Hungary, India, Israel, Mexico, Peru, Poland, Romania, Russia, South Africa, the Ukraine and the United States from 25 June 2008 to 30 August 2010.
Pre-assignment Details: Participants with a historical diagnosis of type 2 diabetes mellitus were enrolled in one of two, once-daily (QD) treatment groups.
Groups:
- Alogliptin 25 mg QD: Alogliptin 25 mg, tablets, orally, once daily and glipizide placebo matching tablets, orally, once daily for up to 52 weeks.
- Glipizide 5 mg QD: Alogliptin placebo-matching tablets, orally, once daily and glipizide 5 mg to 10 mg, tablets, orally, once daily up to 52 weeks.
Period: Overall Study
Arm/Group | Alogliptin 25 mg QD | Glipizide 5 mg QD
Started | 222 | 219
Completed | 133 | 125
Not Completed | 89 | 94
Not completed — Adverse Event | 16 | 20
Not completed — Protocol Violation | 4 | 7
Not completed — Lost to Follow-up | 0 | 4
Not completed — Withdrawal by Subject | 12 | 16
Not completed — Hyperglycemic Rescue | 55 | 47
Not completed — Other | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alogliptin 25 mg QD | Glipizide 5 mg QD | Total
Number analyzed (Participants) | 222 | 219 | 441
Age Continuous [Mean (Standard Deviation); unit: years] | 70.1 (4.42) | 69.8 (4.07) | 69.9 (4.24)
Age, Customized [Number; unit: participants]
  <75 years | 186 | 193 | 379
  ≥75 years | 36 | 26 | 62
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120 | 123 | 243
  Male | 102 | 96 | 198
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 79 | 70 | 149
  Not Hispanic or Latino | 143 | 149 | 292
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 12 | 13 | 25
  Asian | 19 | 26 | 45
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 20 | 36
  White | 169 | 154 | 323
  More than one race | 6 | 6 | 12
  Unknown or Not Reported | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 78.60 (14.842) | 78.81 (15.239) | 78.70 (15.024)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 29.58 (4.348) | 30.02 (4.459) | 29.79 (4.404)
Diabetes duration [Mean (Standard Deviation); unit: years] | 6.25 (6.285) | 5.94 (6.276) | 6.10 (6.275)
Glomerular Filtration Rate (GFR) [Mean (Standard Deviation); unit: mL/min/1.73 m2] — Using the Modification of Diet in Renal Disease method.
  mL/min/1.73 m2 | 73.62 (14.762) | 72.89 (15.524) | 73.26 (15.133)
Smoking history [Number; unit: participants]
  Never smoked | 160 | 168 | 328
  Current smoker | 16 | 11 | 27
  Ex-smoker | 46 | 40 | 86

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin at Week 52.
Description: The change in the percentage of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 52 or final visit and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 52.
Population: Randomized participants who received at least 1 dose of study drug, had measurements at Baseline and at the visit, and who met pre-specified criteria (no major protocol violations) for inclusion in the Per Protocol Set. Missing data were imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 25 mg QD | Glipizide 5 mg QD
Number analyzed (Participants) | 180 | 162
percentage of Glycosylated Hemoglobin | -0.14 (0.063) | -0.09 (0.067)
Statistical Analysis 1: Comparison: Alogliptin 25 mg QD vs Glipizide 5 mg QD; Primary null hypothesis: the average Week 52 HbA1c change from Baseline for alogliptin is inferior to that for glipizide (1-sided 97.5% CI [alpha=0.025] compared to non-inferiority margin of 0.4%). If the primary null hypothesis was rejected (non-inferiority demonstrated), an additional comparison for statistical superiority of alogliptin was performed. The CI was re-evaluated; statistical superiority declared if the upper limit was < 0%; Test type: Superiority or Other; ANCOVA; Treatment, randomization schedule, and geographic region as class effects; baseline value for the endpoint as a continuous covariate; Mean Difference (Final Values) = -0.05, 97.5% CI 1-sided [upper limit 0.13]

2. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at each week indicated including final visit relative to baseline.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, Week 26, Week 34 and Week 42.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 25 mg QD | Glipizide 5 mg QD
Number analyzed (Participants) | 180 | 162
percentage of Glycosylated Hemoglobin
  Week 4 (n=175; n=148) | -0.14 (0.047) | -0.11 (0.051)
  Week 8 (n=180; n=161) | -0.27 (0.051) | -0.23 (0.054)
  Week 12 (n=180; n=162) | -0.34 (0.053) | -0.25 (0.055)
  Week 16 (n=180; n=162) | -0.31 (0.050) | -0.32 (0.052)
  Week 20 (n=180; n=162) | -0.31 (0.051) | -0.27 (0.054)
  Week 26 (n=180; n=162) | -0.28 (0.052) | -0.25 (0.055)
  Week 34 (n=180; n=162) | -0.21 (0.056) | -0.21 (0.059)
  Week 42 (n=180; n=162) | -0.17 (0.062) | -0.17 (0.065)

3. Secondary Outcome: Incidence of Hypoglycemia
Description: Percentage of participants with at least one hypoglycemic episode during 52 week study.
Time Frame: On occurrence (up to 52 weeks).
Population: Percentages based on the number of Safety Set participants in each treatment group.
Measure: Number; unit: percentage of participants
Arm/Group | Alogliptin 25 mg QD | Glipizide 5 mg QD
Number analyzed (Participants) | 222 | 219
percentage of participants | 5.4 | 26.0

4. Secondary Outcome: Incidence of Marked Hyperglycemia (Fasting Plasma Glucose ≥200 mg Per dL).
Description: The number of participants with a fasting plasma glucose value ≥ to 200 mg per dL during the 52 week study.
Time Frame: On Occurrence (up to 52 weeks).
Population: All randomized participants who had at least 1 dose of study medication (full analysis set).
Measure: Number; unit: participants
Arm/Group | Alogliptin 25 mg QD | Glipizide 5 mg QD
Number analyzed (Participants) | 222 | 219
participants
  Baseline to <Week 4 | 30 | 17
  Week 4 to <Week 8 | 11 | 5
  Week 8 to <Week 12 | 12 | 8
  Week 12 to <Week 16 | 11 | 8
  Week 16 to <Week 20 | 5 | 4
  Week 20 to <Week 26 | 2 | 3
  Week 26 to <Week 34 | 3 | 8
  Week 34 to <Week 42 | 2 | 4
  Week 42 to Week 52 | 9 | 6
  Overall | 50 | 37

5. Secondary Outcome: Incidence of Hyperglycemic Rescue
Description: The number of participants requiring rescue for failing to achieve pre-specified glycemic targets during the 52 week study.
Time Frame: On Occurrence (up to 52 weeks).
Population: All randomized participants who had at least 1 dose of study medication (full analysis set). Participants who discontinued prior to Week 2 were excluded from analysis.
Measure: Number; unit: participants
Arm/Group | Alogliptin 25 mg QD | Glipizide 5 mg QD
Number analyzed (Participants) | 222 | 219
participants
  Week 2 to <Week 4 | 1 | 0
  Week 4 to <Week 8 | 2 | 1
  Week 8 to <Week 12 | 1 | 0
  Week 12 to <Week 16 | 14 | 14
  Week 16 to <Week 20 | 6 | 9
  Week 20 to <Week 26 | 5 | 8
  Week 26 to <Week 34 | 10 | 2
  Week 34 to <Week 42 | 6 | 7
  Week 42 to Week 52 | 10 | 6
  Overall | 50 | 37

6. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose
Description: The change in the value of fasting plasma glucose collected at each week indicated including final visit relative to baseline.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, Week 26, Week 34, Week 42 and Week 52.
Population: All randomized participants who had at least 1 dose of study medication (full analysis set) with last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Alogliptin 25 mg QD | Glipizide 5 mg QD
Number analyzed (Participants) | 222 | 219
mg/dL
  Week 2 (n=196; n=199) | -3.8 (1.93) | -5.0 (1.91)
  Week 4 (n=217; n=213) | -7.7 (1.93) | -7.6 (1.95)
  Week 8 (n=217; n=214) | -8.9 (1.76) | -8.7 (1.77)
  Week 12 (n=217; n=214) | -10.2 (1.84) | -9.9 (1.86)
  Week 16 (n=217; n=214) | -7.9 (1.85) | -11.4 (1.86)
  Week 20 (n=217; n=214) | -9.8 (1.78) | -8.7 (1.79)
  Week 26 (n=217; n=214) | -7.9 (1.97) | -6.2 (1.99)
  Week 34 (n=217; n=214) | -5.4 (1.98) | -5.7 (1.99)
  Week 42 (n=217; n=214) | -3.6 (2.13) | -7.4 (2.14)
  Week 52 (n=217; n=214) | -2.4 (2.24) | -4.2 (2.26)

7. Secondary Outcome: Change From Baseline in 2-hour Postprandial Glucose
Description: The change in postprandial (after eating a meal) glucose levels at week 52 relative to baseline. Standard 2-hour postprandial glucose (PPG) tests performed following an overnight fast and evaluated right before and after a 120-minute (2-hour) timeframe relative to ingestion of a standard oral glucose drink.
Time Frame: Baseline and Week 52.
Population: All randomized participants who had at least 1 dose of study medication (full analysis set).
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Alogliptin 25 mg QD | Glipizide 5 mg QD
Number analyzed (Participants) | 222 | 219
mg/dL
  Week 52 PPG level (n=109; n=93) | -5.80 (5.530) | 6.30 (5.989)
  Week 52 PPG excursion (n=109; n=93) | 1.82 (4.434) | 7.17 (4.804)

8. Secondary Outcome: Change From Baseline in Fasting Proinsulin
Description: The change between the value of fasting proinsulin collected at each week indicated including final visit relative to baseline.
Time Frame: Baseline, Week 12, Week 26, Week 42 and Week 52.
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Alogliptin 25 mg QD | Glipizide 5 mg QD
Number analyzed (Participants) | 222 | 219
pmol/L
  Week 12 (n=207; n=186) | -6.0 (0.99) | 1.0 (1.05)
  Week 26 (n=211; n=194) | -4.6 (1.49) | 3.0 (1.56)
  Week 42 (n=211; n=194) | -4.6 (1.48) | 3.1 (1.54)
  Week 52 (n=211; n=194) | -4.9 (1.42) | 3.0 (1.48)

9. Secondary Outcome: Change From Baseline in Insulin
Description: The change between the value of insulin collected at each week indicated including final visit relative to baseline.
Time Frame: Baseline, Week 12, Week 26, Week 42 and Week 52.
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: mcIU/mL
Arm/Group | Alogliptin 25 mg QD | Glipizide 5 mg QD
Number analyzed (Participants) | 222 | 219
mcIU/mL
  Week 12 (n=207; n=188) | -2.36 (0.673) | 0.84 (0.707)
  Week 26 (n=210; n=194) | -0.41 (1.548) | 3.03 (1.611)
  Week 42 (n=210; n=194) | -0.58 (1.254) | 1.53 (1.305)
  Week 52 (n=210; n=194) | -1.72 (1.731) | 3.15 (1.801)

10. Secondary Outcome: Change From Baseline in Proinsulin/Insulin Ratio
Description: The change between the ratio value of proinsulin and insulin collected at each week indicated including final visit relative to baseline.
Time Frame: Baseline, Week 12, Week 26, Week 42 and Week 52.
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Alogliptin 25 mg QD | Glipizide 5 mg QD
Number analyzed (Participants) | 222 | 219
ratio
  Week 12 (n=206; n=185) | -0.288 (0.1035) | 0.053 (0.1092)
  Week 26 (n=210; n=193) | -0.253 (0.4333) | 0.562 (0.4520)
  Week 42 (n=210; n=193) | -0.289 (0.1500) | 0.183 (0.1565)
  Week 52 (n=210; n=193) | -0.155 (0.0899) | -0.057 (0.0938)

11. Secondary Outcome: Homeostasis Model Assessment of Beta Cell Function
Description: The change between homeostasis model assessment of beta cell function collected at each week indicated including final visit relative to baseline. Homeostasis model assessment of beta cell function measures beta cell function, calculated by a constant (20) times insulin, divided by fasting plasma glucose minus a constant (3.5).
Time Frame: Baseline, Week 12, Week 26, Week 42 and Week 52.
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: percent score of beta cell function
Arm/Group | Alogliptin 25 mg QD | Glipizide 5 mg QD
Number analyzed (Participants) | 222 | 219
percent score of beta cell function
  Week 12 (n=203; n=184) | -6.104 (8.3062) | 30.081 (8.7264)
  Week 26 (n=207; n=193) | -0.136 (9.7088) | 31.669 (10.0562)
  Week 42 (n=207; n=193) | -5.571 (7.1395) | 16.004 (7.3950)
  Week 52 (n=207; n=193) | -9.755 (13.8868) | 35.281 (14.3836)

12. Secondary Outcome: Change From Baseline in Body Weight
Description: The change in body weight measured at each week indicated including final visit from baseline.
Time Frame: Baseline, Week 8, Week 12, Week 26, Week 42 and Week 52.
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Alogliptin 25 mg QD | Glipizide 5 mg QD
Number analyzed (Participants) | 222 | 219
kg
  Week 8 (n=213; n=200) | -0.42 (0.118) | 0.55 (0.122)
  Week 12 (n=215; n=203) | -0.52 (0.142) | 0.42 (0.146)
  Week 26 (n=215; n=204) | -0.68 (0.188) | 0.66 (0.193)
  Week 42 (n=215; n=204) | -0.72 (0.211) | 0.57 (0.216)
  Week 52 (n=215; n=204) | -0.62 (0.227) | 0.60 (0.233)

13. Secondary Outcome: Change From Baseline in Serum Lipids (Total Cholesterol)
Description: The change in total cholesterol measured at each week indicated including final visit from baseline.
Time Frame: Baseline, Week 8, Week 12, Week 26, Week 42 and Week 52.
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Alogliptin 25 mg QD | Glipizide 5 mg QD
Number analyzed (Participants) | 222 | 219
mg/dL
  Week 8 (n=208; n=195) | -5.6 (2.01) | -1.6 (2.08)
  Week 12 (n=213; n=201) | -4.2 (2.06) | -0.7 (2.12)
  Week 26 (n=213; n=201) | 1.6 (2.03) | 0.1 (2.09)
  Week 42 (n=213; n=201) | 0.2 (2.07) | 0.1 (2.13)
  Week 52 (n=213; n=201) | -0.8 (2.28) | -0.5 (2.35)

14. Secondary Outcome: Change From Baseline in Serum Lipids (High-Density Lipoprotein Cholesterol)
Description: The change in high-density lipoprotein cholesterol measured at each week indicated including final visit from baseline.
Time Frame: Baseline, Week 8, Week 12, Week 26, Week 42 and Week 52.
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Alogliptin 25 mg QD | Glipizide 5 mg QD
Number analyzed (Participants) | 222 | 219
mg/dL
  Week 8 (n=206; n=193) | -0.1 (0.59) | 1.2 (0.61)
  Week 12 (n=212; n=201) | 0.4 (0.47) | 0.5 (0.48)
  Week 26 (n=212; n=201) | 1.7 (0.50) | 0.2 (0.52)
  Week 42 (n=212; n=201) | 1.4 (0.59) | 0.1 (0.61)
  Week 52 (n=212; n=201) | 0.8 (0.50) | 0.3 (0.51)

15. Secondary Outcome: Change From Baseline in Serum Lipids (Low-Density Lipoprotein Cholesterol)
Description: The change in low-density lipoprotein cholesterol measured at each week indicated including final visit from baseline.
Time Frame: Baseline, Week 8, Week 12, Week 26, Week 42 and Week 52.
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Alogliptin 25 mg QD | Glipizide 5 mg QD
Number analyzed (Participants) | 222 | 219
mg/dL
  Week 8 (n=200; n=185) | -3.2 (1.70) | -2.8 (1.76)
  Week 12 (n=208; n=195) | -2.0 (1.75) | -2.4 (1.81)
  Week 26 (n=208; n=196) | 3.1 (1.67) | -1.1 (1.72)
  Week 42 (n=208; n=197) | 1.2 (1.79) | -0.8 (1.84)
  Week 52 (n=209; n=197) | 0.9 (1.83) | -1.4 (1.88)

16. Secondary Outcome: Change From Baseline in Serum Lipids (Triglycerides)
Description: The change in triglycerides measured at each week indicated including final visit from baseline.
Time Frame: Baseline, Week 8, Week 12, Week 26, Week 42 and Week 52.
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Alogliptin 25 mg QD | Glipizide 5 mg QD
Number analyzed (Participants) | 222 | 219
mg/dL
  Week 8 (n=208; n=195) | -12.8 (5.04) | 2.7 (5.20)
  Week 12 (n=213; n=201) | -15.5 (5.72) | 7.5 (5.89)
  Week 26 (n=213; n=201) | -16.3 (4.74) | 3.9 (4.88)
  Week 42 (n=213; n=201) | -12.6 (5.01) | 5.5 (5.16)
  Week 52 (n=213; n=201) | -13.2 (5.27) | 1.9 (5.42)

17. Secondary Outcome: Change From Baseline in High Sensitivity C-reactive Protein
Description: The change between the high sensitivity C-reactive protein value collected at each week indicated including final visit from baseline.
Time Frame: Baseline, Week 12, Week 26, Week 42 and Week 52.
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: mg/L
Arm/Group | Alogliptin 25 mg QD | Glipizide 5 mg QD
Number analyzed (Participants) | 222 | 219
mg/L
  Week 12 (n=209; n=192) | 0.45 (0.699) | 0.10 (0.730)
  Week 26 (n=212; n=198) | -0.02 (0.682) | 0.47 (0.706)
  Week 42 (n=212; n=198) | 0.33 (0.736) | 0.53 (0.762)
  Week 52 (n=212; n=198) | 0.01 (0.656) | 0.21 (0.679)

18. Secondary Outcome: Incidence of Subjects Achieving Glycosylated Hemoglobin <=7%
Description: The percentage of participants with a value for the percentage of glycosylated hemoglobin (HbA1c; the percentage of hemoglobin that is bound to glucose) less than or equal to 6.5 and 7.0% during the 52 week study.
Time Frame: Baseline and Week 52.
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Alogliptin 25 mg QD | Glipizide 5 mg QD
Number analyzed (Participants) | 222 | 219
percentage of participants
  HbA1c ≤6.5% | 22.3 | 18.2
  HbA1c ≤7.0% | 48.8 | 45.3

19. Secondary Outcome: Incidence of Glycosylated Hemoglobin Decrease From Baseline.
Description: The percentage of participants with a decrease from baseline in the percentage of glycosylated hemoglobin (the percentage of hemoglobin that is bound to glucose) greater than or equal to 0.5, 1.0, 1.5 and 2.0% during the 52 week study.
Time Frame: Baseline and Week 52.
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Alogliptin 25 mg QD | Glipizide 5 mg QD
Number analyzed (Participants) | 222 | 219
percentage of participants
  Decrease from Baseline in HbA1c ≥0.5% | 32.1 | 29.0
  Decrease from Baseline in HbA1c ≥1.0% | 12.6 | 10.3
  Decrease from Baseline in HbA1c ≥1.5% | 5.1 | 2.3
  Decrease from Baseline in HbA1c ≥2.0% | 2.8 | 1.4

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of double-blind study drug and no more than 14 days after the last dose of double-blind study drug.
Description: At each visit the investigator was to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Alogliptin 25 mg QD | Glipizide 5 mg QD
Serious Adverse Events (participants affected / at risk) | 16/222 | 13/219
Other Adverse Events (participants affected / at risk) | 103/222 | 105/219
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alogliptin 25 mg QD (N=222) | Glipizide 5 mg QD (N=219)
Angina pectoris (Cardiac disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 2
Coronary artery disease (Cardiac disorders) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 0
Graft thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1
Left ventricular failure (Cardiac disorders) | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Postoperative fever (Injury, poisoning and procedural complications) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 1 | 0
Stress fracture (Injury, poisoning and procedural complications) | 0 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Urosepsis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alogliptin 25 mg QD (N=222) | Glipizide 5 mg QD (N=219)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 11
Bronchitis (Infections and infestations) | 6 | 9
C-reactive protein increased (Investigations) | 9 | 3
Diarrhoea (Gastrointestinal disorders) | 9 | 14
Dizziness (Nervous system disorders) | 13 | 18
Dyslipidaemia (Metabolism and nutrition disorders) | 5 | 10
Dyspepsia (Gastrointestinal disorders) | 7 | 1
Headache (Nervous system disorders) | 16 | 15
Hypertension (Vascular disorders) | 12 | 10
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 8
Nasopharyngitis (Infections and infestations) | 13 | 10
Nausea (Gastrointestinal disorders) | 7 | 8
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 7
Pharyngitis (Infections and infestations) | 5 | 7
Pyrexia (General disorders) | 2 | 7
Upper respiratory tract infection (Infections and infestations) | 12 | 5
Urinary tract infection (Infections and infestations) | 26 | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be published prior to publication of a multi-center report submitted for publication within 18 months after conclusion or termination of a study at all study sites. Results publications will be submitted to sponsor for review 60 days in advance of publication. Sponsor can require removal of confidential information unrelated to study results. Sponsor can embargo a proposed publication for another 60 days to preserve intellectual property.